CLINICAL TRIAL: NCT04212910
Title: Stratifying Endometrial Cancer Patients Using a PET/MRI Prognostic Model
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco De Cobelli, Head, Radiology Department, IRCCS San Raffaele
Other Study IDs: PET/MRI-ONCOGYN
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Endometrium Cancer
Keywords: endometrium; cancer; PET-MRI; stratification
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Surgically removed endometrium and lymphnodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial cancer (EC) is the most common gynecological malignancy in high-income countries. Prognosis and treatment are dictated by cancer histological subtype and grade coupled with surgical staging as described by Surgical International Federation of Gynecology and Obstetrics (FIGO) staging system. Surgery is the elective standard treatment and used for staging of EC. The purpose of this study is to collect images from a simultaneous PET/MRI study from which to extrapolate a preoperative, non-invasive, prognostic model.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is the most frequently used imaging tool in preoperative staging of endometrial cancer. FDG-PET has demonstrated higher sensitivity than MRI in detecting nodal involvement and metastatic disease and is currently used in adjunction to MRI. Distinct MRI and FDG-PET parameters correlate well with tumor aggressiveness and can and have been used as prognostic factors. The Investigators believe that the combination of data from these two imaging techniques, from which different derived tumor features can be extrapolated, can stratify patients in high-risk and low-risk groups already preoperatively. The aim of combined techniques is to collect large amounts of data leveraging advantages of both modalities (MR's strengths in local staging and PET's strengths in nodal staging) in a single scan from which to extrapolate a preoperative, non-invasive, prognostic model.

ELIGIBILITY:
Inclusion Criteria:

* histopathological confirmation of a primary endometrial cancer
* age > 18 years
* no contraindication to surgery (comorbidity, contraindication or lack of consent)
* no contraindication to preoperative imaging
* visible tumor at imaging
* signed inform consent.

Exclusion Criteria:

* patients unsuitable for surgical intervention (comorbidity, contraindication or lack of consent, poor performance status)
* age < 18 years, c) inability to complete the needed imaging examination (ie, severe claustrophobia)
* any additional medical condition that may significantly interfere with study compliance
* all the contraindication for MRI (ie, pacemaker).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females patients with endometrial cancer
Study Population: Patients with biopsy proven endometrial cancer presenting to the Institution's Gynecology Unit.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
MRI evaluation | 0-2 years
  Measure tumor volume and correlate to surgical specimen
MRI imaging | 0-2 years
  Changes in ADC normale versus tumor myometrium
MRI imaging evaluation | 0-2 years
  Depth of myometrial invasion
DCE-MRI perfusion parameters | 0-2 years
  Define tumor perfusion in normal versus tumor myometrium
MRI | 0-2 years
  positive lymph node evaluation
PET imaging evaluation | 0-2 years
  PET positive lymph nodes
PET imaging | 0-2 years
  Tumor/positive lymph node/metastases SUV values

SECONDARY OUTCOMES:
Measure tumor angiogenesis | 0-2 years
  angiogenesis marker, CD1
Correlate PET and MRI derived functional and morphological parameters with histology | 0-5 years
  Imaging derived parameters correlated with histopathology

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitajima K, Kita M, Suzuki K, Senda M, Nakamoto Y, Sugimura K. Prognostic significance of SUVmax (maximum standardized uptake value) measured by [(1)(8)F]FDG PET/CT in endometrial cancer. Eur J Nucl Med Mol Imaging. 2012 May;39(5):840-5. doi: 10.1007/s00259-011-2057-9. Epub 2012 Feb 17. PMID 22349717
- [Background] Nakamura K, Kodama J, Okumura Y, Hongo A, Kanazawa S, Hiramatsu Y. The SUVmax of 18F-FDG PET correlates with histological grade in endometrial cancer. Int J Gynecol Cancer. 2010 Jan;20(1):110-5. doi: 10.1111/IGC.0b013e3181c3a288. PMID 20130510
- [Derived] Bezzi C, Ironi G, Russo T, Candotti G, Fallanca F, Sabini C, Samanes Gajate AM, Ghezzo S, Bergamini A, Sant'Angelo M, Bocciolone L, Brembilla G, Scifo P, Taccagni G, Catalano OA, Mangili G, Candiani M, De Cobelli F, Chiti A, Mapelli P, Picchio M. [18F]FDG PET/MRI in Endometrial Cancer: Prospective Evaluation of Preoperative Staging, Molecular Characterization and Prognostic Assessment. Cancers (Basel). 2026 Jan 16;18(2):280. doi: 10.3390/cancers18020280. PMID 41595203